CLINICAL TRIAL: NCT06107777
Title: The Efficacy of Pharmacopuncture on Inpatients With Psychological Stress Caused by Traffic Accidents: A Practical Randomized Control Pilot Study
Brief Title: The Effectiveness of Pharmacopuncture on Psychological Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jaseng Medical Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JS-CT-2023-05
Record Dates: First submitted 2023-10-12; First posted 2023-10-30 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-03

CONDITIONS: Psychological Stress
Keywords: Psychological Stress; Pharmacopuncture
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pharmacopucture on Acupoints Related to Psychological Stress (Experimental): The Pharmacopucture group will recieve Pharmacopucture treatment durling the hospitalization. The mandatory acupoints are (Dan-jung(CV17), Jung-wan(CV12), Gi-hae(CV6), Gwan-won(CV4), Sin-mun(HT7). If needed, they will recieve additional acupoints are (So-hae(HT3), Jung-jeo(TE3), Sam-eumgyo(SP6). A trained doctor of Korean medicine with at least 3 years of clinical experience are going to conduct the pharmacopucture.
  The Pharmacopucture group will also be treated with other Korean medical treatment everyday: acupuncture, chuna and Korean herbal medicine.
  Interventions: Procedure: Pharmacopuncture; Procedure: Korean medical treatment
- Korean medical treatment (Active Comparator): The control group will receive Korean medical treatment everyday after hospitalization: acupuncture, chuna, pharmacoacupuncture(except on mandatory and additional acupoints) and Korean herbal medicine.
  Interventions: Procedure: Korean medical treatment

INTERVENTIONS:
Procedure: Pharmacopuncture — Pharmacopuncture is a treatment that combines 2 of the most frequented Korean medicine treatment methods - traditional acupuncture and herbal medicine - by injecting herbal medicine extract at acupoints.
  Arms: Pharmacopucture on Acupoints Related to Psychological Stress
Procedure: Korean medical treatment — acupuncture treatment, chuna, pharmacoacupuncture, Korean herbal medicine

SUMMARY:
This study is a double blind, randomized controlled trail. Condition/disease: Psychological Stress treatment Intervention:Pharmacopuncture

DETAILED DESCRIPTION:
"Pharmacopuncture is a treatment that combines 2 of the most frequented Korean medicine treatment methods - traditional acupuncture and herbal medicine - by injecting herbal medicine extract at acupoints.

This treatment is known to be an important part of Korean medicine treatment. However, there has been no specific value for the effect of this treatment.

Therefore, the investigators are going to conduct a practical randomized controlled trials to verify the efficacy and safety of Pharmacopuncture on Psychological Stress. From October 2023 to December 2024, the investigators are going to collect 50 inpatients who are suffering from Psychological Stress with the HADS-A(Hospital Anxiety and Depression Scale-anxiety) or HADS-D(Hospital Anxiety and Depression Scale-Depression) over 8 after injury by traffic accident(TA). For experimental group(n=25), the investigators will conduct Pharamacopuncture on 5 mandatory acupoints and 3 additional acupoints if needed durling the hospitalization and other Korean medical treatment. For control group(n=25), just Korean medical treatment except Pharamacopuncture on mandatory acupoints and additional acupoints will be conducted.

For these two groups, the investigators will compare Psychological stress intensity scale: Hospital Anxiety and Depression Scale (HADS), NRS of Anxiety, NRS of Depression, NRS of Physical pain, Sleeping disorder intensity scale: Korean version of the Insomnia Severity Index(ISI-K), subjective stress scale caused by traumatic events: Revised Version of the Impact of Event Scale of Korea(IES-R-K), EuroQol 5-Dimension (EQ-5D-5L) and Patient Global Impression of Change (PGIC)."

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 19-69 years on the date they sign the consent form.
* Patients who are suffered by Psychological Stress that occurred within 3 days after traffic accident.
* Patients who are hospitalized due to traffic accident.
* Patients with HADS-A ≥ 8 or HADS-D ≥ 8.
* Patients who provide consent to participate in the trial and return the informed consent form.

Exclusion Criteria:

* Patients with progressive neurological deficit or with serious neurological symptoms.
* Patients with a specific serious disease that may interfere with the interpretation of the therapeutic effects or results: malignancy, spondylitis, inflammatory spondylitis, etc.
* Patients who are taking steroids, immunosuppressants, mental illness drugs, or other drugs that may affect the results of the study.
* Patients with medical history of brain disease or surgery due to trauma.
* Patients who are addicted by drug or alcohol within the year.
* If acupuncture is inadequate or unsafe: patients with hemorrhagic, receiving anticoagulants, severe diabetes and cardiovascular disease.
* Patients who are pregnant or planning to become pregnant
* Patients who are participated in clinical trials other than observational studies without therapeutic intervention.
* Patients who are difficult to complete the research participation agreement
* Other patients whose participation in the trial is judged by a researcher to be problematic

Ages: 19 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-11-20 (Actual); Primary Completion 2024-06-26 (Actual); Study Completion 2024-06-26 (Actual)

PRIMARY OUTCOMES:
Hospital Anxiety and Depression Scale(HADS) | Screeing day (day 1), Baseline (day2), Discharge 1 day, 15 days after admission day, 2 months after admission day
  Hospital Anxiety and Depression Scale aims to measure symptoms of anxiety and depression. It is a self-rating scale developed to assess psychological distress in non-psychiatric patients. The HADS consists of 14 questions and each question is scored on a 4-point Likert scale(0=no problems, 3=severe problems) The odd numbers ask anxiety(HADS-A) and even number ask Depression(HADS-D). HADS-A (or HADS-D) cut-off score is 8 or above.

SECONDARY OUTCOMES:
Korean version of the Insomnia Severity Index(IES-R-K) | Baseline (day2), Discharge 1 day, 15 days after admission day, 2 months after admission day
  IES-R-K is the Korean version of impact of event scale revised. It was designed as a measure of post-traumatic stress disorder (PTSD) symptoms, and is a short, easily administered self-report questionnaire. It has 22 items and a cut-off score of 33 or above.
Korean version of the Insomnia Severity Index(ISI-K) | Baseline (day2), Discharge 1 day, 15 days after admission day, 2 months after admission day
  ISI-K is a Korean version of Insomnia Severity Index. It was designed as a brief screening tool for insomnia and has the seven-item questionnaire asks respondents to rate the nature and symptoms of their sleep problems using a Likert-type scale.
Numeric Rating Scale of Anxiety (NRS of Anxiety) | From baseline(Day2) up to Discharge 1 day, 15 days after admission day, 2 months after admission day
  NRS is a pain scale in which the patient indicates their subjective pain as a whole number from 0 to 10. The participant is asked to report their Anxiety using NRS, where 0 indicates 'no pain or discomfort' and 10 indicates 'the most severe pain and discomfort imaginable'.
Numeric Rating Scale of Depression(NRS of Depression) | From baseline(Day2) up to Discharge 1 day, Discharge 1 day, 15 days after admission day, 2 months after admission day
  NRS is a pain scale in which the patient indicates their subjective pain as a whole number from 0 to 10. The participant is asked to report their Depression using NRS, where 0 indicates 'no pain or discomfort' and 10 indicates 'the most severe pain and discomfort imaginable'.
Numeric Rating Scale of Physical pain(NRS of Physical pain) | From baseline(Day2) up to Discharge 1 day, Discharge 1 day, 15 days after admission day, 2 months after admission day
  NRS is a pain scale in which the patient indicates their subjective pain as a whole number from 0 to 10. The participant is asked to report their Physical pain and discomfort using NRS, where 0 indicates 'no pain or discomfort' and 10 indicates 'the most severe pain and discomfort imaginable'.
EuroQol 5-Dimension (EQ-5D) | Baseline(day2), Discharge 1 day, 15 days after admission day, 2 months after admission day
  The EQ-5D is a method of indirectly calculating the weights of certain health states for quality of life after a multidimensional investigation of health states, and is the most widely used instrument for this purpose. The EQ-5D consists of 5 questions about current health state (mobility, self-care, usual activities, pain, anxiety/depression), and each question is scored on a 5-point Likert scale (1=no problems, 3=moderate problems, 5=severe problems). In this study, the investigators will use the Korean version of the EQ-5D, which has been demonstrated to be valid.
Patient Global Impression of Change (PGIC) | Discharge 1 day, 15 days after admission day, 2 months after admission day
  The PGIC is an index that assesses improvements in functional limitation caused by whiplash injury. Participants rate the improvement in functional limitations after treatment on a 7-point Likert scale (1=Very much improved, 4=No change, 7=Very much worse). This index was originally developed for use in Psychology, but is currently used in various other medical fields to assess improvements in pain.

CONTACTS AND LOCATIONS:
Overall Officials: In-Hyuk Ha, phD, Principal Investigator — Jaseng Medical Foundation
Locations (1):
- Jaseng Hospital of Korean Medicine, Seoul, Gangnam-Gu, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Son JY, Jung S, Lee YH, Kim DG, Kim JW, Lee TJ, Cho SH, Ji JH, Cho HW, Kim SD, Lee YJ, Ha IH, Kim D, Shin BC. Pharmacopuncture for patients with psychological stress caused by traffic accidents: A pragmatic randomized controlled pilot trial. Integr Med Res. 2026 Mar;15(1):101251. doi: 10.1016/j.imr.2025.101251. Epub 2025 Sep 1. PMID 40995057